CLINICAL TRIAL: NCT02815475
Title: Turmeric Anti-Inflammatory and Cell-Damage Trial
Acronym: TACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Collaborators: British Broadcasting Corporation (Industry); University College, London (Other); University of Leeds (Other); PB Biosystems Ltd (Unknown)
Responsible Party: Principal Investigator, Anthony Watson, Research Associate, Newcastle University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NUHEALTH-KB01-TACT
Record Dates: First submitted 2016-06-20; First posted 2016-06-28 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Starch filled capsule
  Interventions: Dietary Supplement: Placebo comparator
- Curcumin (Experimental): 400mg of Curcumin via capsule to be consumed every other day
  Interventions: Dietary Supplement: Curcumin
- Turmeric powder (Active Comparator): 2 teaspoons of dried turmeric powder to be consumed every other day
  Interventions: Dietary Supplement: Turmeric powder

INTERVENTIONS:
Dietary Supplement: Placebo comparator
  Arms: Placebo
Dietary Supplement: Curcumin
  Arms: Curcumin
Dietary Supplement: Turmeric powder
  Arms: Turmeric powder

SUMMARY:
This trial will be conducted for the BBC. The aim of the project is to assess if consuming the spice turmeric every other day, in the amount consumed in a curry, can reduce cell damage and inflammation. The results of the project will be used to inform the TV program Trust Me I'm a Doctor.

DETAILED DESCRIPTION:
100 volunteers will be recruited for a 6 week intervention. The study group will be divided into 3 arms, each with approximately. 33 participants; one arm will receive a placebo capsule, one arm will receive a capsule with 400mg of curcumin (corresponding to two teaspoons of turmeric powder). These treatments are done double-blind. A third arm is 'open label', these volunteers will receive a bag with at least 135g turmeric and be asked to add two teaspoon to their food. Participants will be asked to supplement their diet with turmeric (powder, capsule or placebo) every other day for six weeks.

Participants will be asked to attend the NU-Food research facility on 3 occasions. The first will be a screening session where participants will be given the option to discuss the project with a researcher. Participants will complete a screening questionnaire and sign an informed consent form. On the next visit, participants will arrive at the research facility at a pre-arranged time and firstly have their height and weight measured. Participants will then give 10ml of blood via venepuncture and asked to provide a 10ml spot urine sample. After this participants will be randomly allocated a treatment group (placebo, turmeric capsule or turmeric powder) and given instructions on dosage. After a 6 week treatment period, participants will return to the research facility, have their height and weight measured then give a second 10ml venous blood sample and provide a final spot urine sample. Each visit will take around 20 minutes.

The main outcomes of the trial are oxidative stress and inflammation tests which will be conducted by PB bioscience and an assessment of DNA methylation by University College London. Proteomics analysis will be conducted on Urine samples.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and over
* No pre-existing medical conditions
* not currently taking prescribed drugs or over the counter supplements
* Male and female

Exclusion Criteria:

* Any pre-existing medical condition
* Taking prescribed drugs or over the counter supplements
* Aged 17 years or under
* BMI > 40mg/m2
* BP > 160/120

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline DNA methylation analyses based on the Illumina EPIC array | Baseline and 6 weeks post dose
Change from baseline oxidative stress determination using whole-blood chemiluminescence assays | Baseline and 6 weeks post dose

CONTACTS AND LOCATIONS:
Locations (1):
- NU-Food, Newcastle upon Tyne, Tyne and Wear, United Kingdom